CLINICAL TRIAL: NCT03849690
Title: A Single-Sequence, Open-Label, 2-Period, Crossover Trial to Evaluate the Effect of the Proton Pump Inhibitor Esomeprazole on the Single-Dose Pharmacokinetics of Oral TAK-906 in Healthy Adult Subjects
Brief Title: A Trial to Evaluate the Effect of the Proton Pump Inhibitor Esomeprazole on the Single-dose Pharmacokinetics (PK) of Oral TAK-906 in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TAK-906-1006; U1111-1224-9867 (Registry Identifier: WHO)
Record Dates: First submitted 2019-02-20; First posted 2019-02-21 (Actual); Results first posted 2020-05-12 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-05

CONDITIONS: Healthy Volunteers
Keywords: Drug Therapy
MeSH Terms: interventions — trazpiroben; Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TAK-906 25 mg; Esomeprazole 40 mg + TAK-906 25 mg (Experimental): TAK-906 25 milligram (mg), capsule, orally, once on Day 1 of Study Period 1, followed by a washout period of at least 4 days, further followed by esomeprazole 40 mg, capsule, orally, once daily on Days 1 to 5 along with TAK-906 25 mg, capsule, orally, once on Day 4 of Study Period 2.
  Interventions: Drug: TAK-906; Drug: Esomeprazole

INTERVENTIONS:
Drug: TAK-906 — TAK-906 capsules.
  Other Names: TAK-906 maleate
Drug: Esomeprazole — Esomeprazole capsules.
  Other Names: Nexium

SUMMARY:
The purpose of this study is to evaluate the effect of the proton pump inhibitor (PPI) esomeprazole on the single-dose PK of orally administered TAK-906.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-906. TAK-906 is being tested in healthy participants to evaluate the effect of a PPI esomeprazole on the PK of TAK-906.

The study will enroll approximately 12 participants. Participants will be assigned to the following treatment sequence:

• TAK-906 25 mg; Esomeprazole 40 mg + TAK-906 25 mg

All participants will be given an oral dose of TAK-906 and Esomeprazole.

This single center trial will be conducted in the United States. The overall duration to participate in this study is 52 days. Participants will make visit to the clinic during Period 1 and Period 2 in addition to approximately 10 to 14 days after receiving their last dose of TAK-906 for a follow up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Continuous non-smoker who has not used nicotine containing products for at least 3 months prior to the first dosing and throughout the study, based on screening urine cotinine test.
2. Has a body mass index (BMI) greater than or equal to (>=) 18 and less than or equal to (<=) 30 kilogram per square meter (kg/m^2) at Screening.

Exclusion Criteria:

1. History or presence of alcoholism or drug abuse within the past 2 years prior to the first dosing.
2. QT interval corrected using Fridericia's formula (QTcF) interval is greater than (>) 450 millisecond (msec) or ECG findings are deemed abnormal with clinical significance by the Investigator or designee at screening.
3. Donation of blood or significant blood loss (example, approximately 500 milliliter [mL]) within 56 days prior to the first dosing.
4. Plasma donation within 7 days prior to the first dosing.
5. Participation in another clinical study within 30 days or 5 half-lives prior to the first dosing. The 30 day window or 5 half-lives will be derived from the date of the last blood collection or dosing, whichever is later, in the previous study to Day 1 of Study Period 1 of the current study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2019-02-27 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Millennium Pharmaceuticals, Inc.
Locations (1):
- Celerion, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Kaur Mukker J, Dukes G, Wang L, Huh S, Khudyakov P, Nishihara M, Chen C. Evaluation of the pharmacokinetics of trazpiroben (TAK-906) in the presence and absence of the proton pump inhibitor esomeprazole. Clin Transl Sci. 2022 May;15(5):1281-1290. doi: 10.1111/cts.13248. Epub 2022 Feb 26. PMID 35218604

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in the Unites states from 27 February 2019 to 15 April 2019.
Pre-assignment Details: Healthy participants were enrolled in this single sequence, 2-period cross-over design study to receive TAK-906 25 milligram (mg) in Study Period 1 followed by esomeprazole 40 mg and TAK-906 25 mg in Study Period 2.
Groups:
- TAK-906 25 mg + Esomeprazole 40 mg and TAK-906 25 mg: TAK-906 25 mg, capsule, orally, once on Day 1 of Study Period 1, followed by a washout period of at least 4 days, further followed by esomeprazole 40 mg, capsule, orally, once daily on Days 1 to 5 along with TAK-906 25 mg, capsule, orally, once on Day 4 of Study Period 2.
Period: Period 1 (3 Days)
Arm/Group | TAK-906 25 mg + Esomeprazole 40 mg and TAK-906 25 mg
Started | 12
Completed | 12
Not Completed | 0
Period: Washout Period (at Least 4 Days)
Arm/Group | TAK-906 25 mg + Esomeprazole 40 mg and TAK-906 25 mg
Started | 12
Completed | 12
Not Completed | 0
Period: Period 2 (6 Days)
Arm/Group | TAK-906 25 mg + Esomeprazole 40 mg and TAK-906 25 mg
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The safety set included all participants who received at least one dose of study drug.
Arm/Group | TAK-906 25 mg + Esomeprazole 40 mg and TAK-906 25 mg
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.8 (9.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 72.30 (11.532)
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 168.5 (8.48)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 25.315 (2.4635)

OUTCOME MEASURES:

1. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-906
Time Frame: TAK-906 25 mg: Day 1 pre-dose and at multiple time points (up to 48 hours) post-TAK-906 dose; Esomeprazole 40 mg and TAK-906 25 mg: Day 4 pre-dose and at multiple time points (up to 48 hours) post-TAK-906 dose
Population: The pharmacokinetic (PK) set included all participants who complied sufficiently with the protocol and displayed an evaluable PK profile (example, exposure to treatment, availability of measurements and absence of major protocol violations).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Groups:
- TAK-906 25 mg: TAK-906 25 mg, capsule, orally, once on Day 1 of Study Period 1.
- Esomeprazole 40 mg and TAK-906 25 mg: Esomeprazole 40 mg, capsule, orally, once daily on Days 1 to 5 along with TAK-906 25 mg, capsule, orally, once on Day 4 of Study Period 2.
Arm/Group | TAK-906 25 mg | Esomeprazole 40 mg and TAK-906 25 mg
Number analyzed (Participants) | 12 | 12
nanogram per milliliter (ng/mL) | 19.76 (36.5) | 17.24 (40.5)
Statistical Analysis 1: Comparison: TAK-906 25 mg vs Esomeprazole 40 mg and TAK-906 25 mg; Test type: Other — Analysis of variance (ANOVA) performed on natural log(ln)-transformed TAK-906 Cmax which exponentiated to provide estimates on original scale. ANOVA model included treatment as fixed effect and participant as random effect. Each ANOVA included calculation of least-squares means(LSM) and difference between treatment LSM. Geometric mean ratios and 90% confidence interval (CI) were determined by exponentiation of appropriate estimates for difference between treatments in log-transformed parameters; p = 0.3011, ANOVA; Geometric mean ratio = 0.87, 90% CI 2-sided [0.70 to 1.09]

2. Primary Outcome: AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for TAK-906
Time Frame: TAK-906 25 mg: Day 1 pre-dose and at multiple time points (up to 48 hours) post-TAK-906 dose; Esomeprazole 40 mg and TAK-906 25 mg: Day 4 pre-dose and at multiple time points (up to 48 hours) post- TAK-906 dose
Population: The PK set included all participants who complied sufficiently with the protocol and displayed an evaluable PK profile (example, exposure to treatment, availability of measurements and absence of major protocol violations).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*h/mL)
Arm/Group | TAK-906 25 mg | Esomeprazole 40 mg and TAK-906 25 mg
Number analyzed (Participants) | 12 | 12
nanogram*hour per milliliter (ng*h/mL) | 43.31 (27.8) | 37.98 (31.2)
Statistical Analysis 1: Comparison: TAK-906 25 mg vs Esomeprazole 40 mg and TAK-906 25 mg; Test type: Other — ANOVA was performed on ln-transformed TAK-906 AUClast which were exponentiated to provide estimates on original scale. ANOVA model included treatment as fixed effect and participant as a random effect. Each ANOVA included calculation of LSM and difference between treatment LSM. Geometric mean ratios and 90 percent (%) CI were determined by exponentiation of appropriate estimates for difference between treatments in log-transformed parameters; p = 0.0865, ANOVA; Geometric mean ratio = 0.88, 90% CI 2-sided [0.77 to 0.99]

3. Primary Outcome: AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-906
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | TAK-906 25 mg | Esomeprazole 40 mg and TAK-906 25 mg
Number analyzed (Participants) | 12 | 12
ng*h/mL | 44.03 (27.5) | 38.85 (31.1)
Statistical Analysis 1: Comparison: TAK-906 25 mg vs Esomeprazole 40 mg and TAK-906 25 mg; Test type: Other — ANOVA was performed on ln-transformed TAK-906 AUC∞ which were exponentiated to provide estimates on original scale. ANOVA model included treatment as fixed effect and participant as a random effect. Each ANOVA included calculation of LSM and difference between treatment LSM. Geometric mean ratios and 90% CI were determined by exponentiation of appropriate estimates for difference between treatments in log-transformed parameters; p = 0.3011, ANOVA; Geometric mean ratio = 0.88, 90% CI 2-sided [0.78 to 1.00]

4. Secondary Outcome: Number of Participants Who Experienced at Least One Treatment Emergent Adverse Event (TEAE), Serious Adverse Event (SAE), and Grade 3 or Higher TEAEs
Description: A severity grade is defined by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 5.0. Grade 1 scales as Mild (asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated); Grade 2 scales as Moderate (minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental ADL); Grade 3 scales as severe(severe or medically significant but not immediately life threatening hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL); Grade 4 scales as life-threatening consequences, urgent intervention indicated, and Grade 5 scales as death related to AE.
Time Frame: Baseline up to 14 days after last dose of TAK-906 in Study Period 2 (Day 23)
Population: The safety set included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Esomeprazole 40 mg: Esomeprazole 40 mg, capsule, orally, once daily on Days 1 to 5 of Study Period 2.
Arm/Group | TAK-906 25 mg | Esomeprazole 40 mg | Esomeprazole 40 mg and TAK-906 25 mg
Number analyzed (Participants) | 12 | 12 | 12
Participants
  TEAEs | 2 | 1 | 3
  SAEs | 0 | 0 | 0
  Grade 3 or Higher TEAEs | 0 | 0 | 0

5. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in Vital Signs
Time Frame: Baseline up to 14 days after last dose of TAK-906 in Study Period 2 (Day 23)
Population: The safety set included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | TAK-906 25 mg | Esomeprazole 40 mg | Esomeprazole 40 mg and TAK-906 25 mg
Number analyzed (Participants) | 12 | 12 | 12
Participants | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in 12-lead Electrocardiogram (ECG)
Time Frame: Baseline up to 14 days after last dose of TAK-906 in Study Period 2 (Day 23)
Population: The safety set included all participants who received at least one dose of study drug. The safety set where data at specified time points was available.
Measure: Count of Participants; unit: Participants
Arm/Group | TAK-906 25 mg | Esomeprazole 40 mg | Esomeprazole 40 mg and TAK-906 25 mg
Number analyzed (Participants) | 12 | 12 | 12
Participants | 0 | 0 | 0

7. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline Clinical Laboratory Values
Time Frame: Baseline up to 14 days after last dose of TAK-906 in Study Period 2 (Day 23)
Population: The safety set included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | TAK-906 25 mg | Esomeprazole 40 mg | Esomeprazole 40 mg and TAK-906 25 mg
Number analyzed (Participants) | 12 | 12 | 12
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: TEAEs are AEs that started after the first dose of study drug and no more than 14 days after the last dose of study drug in Study Period 2 (Day 23)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | TAK-906 25 mg | Esomeprazole 40 mg | Esomeprazole 40 mg and TAK-906 25 mg
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 2/12 | 1/12 | 3/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TAK-906 25 mg (N=12) | Esomeprazole 40 mg (N=12) | Esomeprazole 40 mg and TAK-906 25 mg (N=12)
Influenza like illness (General disorders) | 0 | 0 | 1
Vessel puncture site pain (General disorders) | 0 | 0 | 1
Vessel puncture site reaction (General disorders) | 0 | 0 | 1
Folliculitis (Infections and infestations) | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 0
Menstruation delayed (Reproductive system and breast disorders) | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2019-02-04): https://cdn.clinicaltrials.gov/large-docs/90/NCT03849690/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-22): https://cdn.clinicaltrials.gov/large-docs/90/NCT03849690/SAP_001.pdf